CLINICAL TRIAL: NCT05819177
Title: An Analysis of the Information of the Coma Recovery Scale-Revised Providing the Most Reliable Prediction of the Neurobehavioral State and Recovery of Consciousness
Brief Title: Information of the Coma Recovery Scale-Revised for Neurobehavioral State and Recovery of Consciousness Prediction
Acronym: CRS-R_Info
Status: Completed | Type: Observational
Sponsor: Hospitales Nisa (Other)
Responsible Party: Sponsor
Other Study IDs: CRS-R_Info
Record Dates: First submitted 2023-03-09; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Disorder of Consciousness
Keywords: Disorders of consciousness; Unresponsive wakefulness syndrome; Minimally conscious state; Severe brain injury; Prognosis; Machine learning
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort undergoing rehabilitation: This group of patients underwent standard rehabilitation programs set by national guidelines.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — This group of patients underwent standard rehabilitation programs set by national guidelines.

SUMMARY:
Background: The Coma Recovery Scale-Revised (CRS-R) is the most recommended instrument to examine the neurobehavioral condition of individuals with disorders of consciousness (DOCs). Different studies have investigated the prognostic value of the information provided by the conventional administration of the scale, while other measures derived from the scale have been proposed to improve the prognosis of DOCs. However, the heterogeneity of the data used in the different studies prevents a reliable comparison of the identified predictors and measures.

Objectives: This study investigates which information derived from the CRS-R provides the most reliable prediction of both the neurobehavioral state and recovery of consciousness at the discharge of a long-term neurorehabilitation program.

Methods: The clinical records of 171 individuals with DOCs admitted to an inpatient neurorehabilitation program for a minimum of 3 months were used to implement machine learning classifiers that were trained to predict the neurobehavioral state and recovery of consciousness at discharge.

DETAILED DESCRIPTION:
Severe acquired brain injury, understood as any damage to the brain that causes coma for over 24 hours, can lead to a complex clinical condition characterized by impaired consciousness, commonly referred to as a disorder of consciousness (DOC). The concept of consciousness is multifaceted and complex and arises from the presence of both arousal, i.e. vigilance and wakefulness, and awareness, i.e. perception of the environment and self. Consequently, depending on the presence and nature of the behavioral responses to multisensory stimuli, individuals with DOC are diagnosed as either in an unresponsive wakefulness syndrome (UWS) or vegetative state (VS) if they only show reflexes, or in a minimally conscious state (MCS) if they show intentional responses. Two further subgroups have been proposed within this latter group that allow to categorize individuals in an MCS+ or in an MCS- according to the presence or absence of higher-level behaviors, respectively. Finally, individuals who show functional communication or functional use of objects are considered as emerging from the MCS.

Diagnosis of DOCs, therefore, poses a clinical challenge, as it requires the accurate analysis of behavioral signs that can be weak or inconsistent. The Coma Recovery Scale-Revised (CRS-R) is the most recommended instrument worldwide for assessing the neurobehavioral condition of individuals with DOC and features multiple cross-cultural adaptations. The CRS-R investigates the presence of 23 neurobehavioral responses, grouped in 6 different subscales, which evaluate auditory, visual, motor, oromotor, communication, and arousal functions. For each subscale, the responses are hierarchically ordered and are evaluated from higher responses (cognitively-mediated responses) to lower responses (reflexes). The diagnostic utility of the scale was first analyzed in 2004, but it was not until 2010 that its interrater reliability, internal consistency, and prognostic or diagnostic validity supported its use for diagnosis. Additionally, although this has been only proven for traumatic etiology, the scale has demonstrated strong construct validity, with confirmed evidence of monotonicity, mutual independence, and invariant item ordering. In this regard, the hierarchy of the CRS-R has also shown a lack of invariance across relevant group factors including age, sex, etiology, enrollment facility, time since injury, and time between assessments. However, in spite that all these properties of the CRS-R contribute to reduce its diagnostic error in comparison to consensus-based tools, it is recommended that the diagnosis of DOCs is based on the clinical findings from five consecutive assessments and combined with imaging or electrophysiological-derived measures. Interestingly, some authors have proposed alternative indices and measures derived from the CRS-R, such as the CRS-R Modified Score and the CRS-R Index, pursuing an increase in the accuracy of the original version.

The total score in the CRS-R has been also identified as an important predictor of recovery of responsiveness in non-traumatic individuals with UWS in Class I studies. In the case of mixed cohorts, however, the current guidelines neither confirm nor refuse the prognostic value of the CRS-R due to insufficient evidence. However, more recent studies highlight the relevance of the information provided by the CRS-R in the prediction of the recovery of consciousness. Measures derived from the CRS-R have been also proposed to improve prognosis of DOCs. Arnaldi and colleagues introduced the CRS+, a weighted score based on the CRS-R to investigate the prognostic value of sleep patterns in the recovery of consciousness. More recently, the Consciousness Domain Index was proposed, an unsupervised machine learning clustering technique based on information from the CRS-R sub-scales to improve the prediction of recovery of consciousness.

However, although the information provided by the CRS-R might be essential to predict the clinical progress of individuals with DOCs and many attempts exist to find alternative measures that improve the predictive value of the original instrument, the heterogeneity of the data used in the different studies prevent a reliable comparison of the identified predictors and measures. Consequently, the aim of this study was to determine which information derived from the CRS-R provides the most reliable prediction of both the neurobehavioral state and recovery of consciousness at discharge of a long-term neurorehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with (Unresponsive Wakefulness Syndrome) UWS or Minimal Consciousness State (MCS) due to either a vascular, anoxic or traumatic origin

Exclusion Criteria:

* individuals who did not attended the program for at least three months

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Disorder Of Consciousness (DOC) who had attended an inpatient neurorehabilitation program between February 2004 and December 2021 in three facilities of the same hospital network were retrospectively extracted from their medical records.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2004-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recovery of consciousness | At discharge from the rehabilitation hospital (median of 365 days)
  Described as Emergence from Minimal Consciousness State (MCS) or from Unresponsive Wakefulness Syndrome (UWS) (1) or presence of Disorder of Consciousness (DoC, 0)
Neurobehavioral state | At discharge from the rehabilitation hospital (median of 365 days)
  Described as Minimal Consciousness State (MCS), Unresponsive Wakefulness Syndrome (UWS), or Emergence from Minimal Consciousness State (E-MCS)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospitales NISA, Valencia
  - Servicio de Neurorrehabilitación y Daño Cerebral de los Hospitales NISA, Valencia

REFERENCES:
- [Background] Hirschberg R, Giacino JT. The vegetative and minimally conscious states: diagnosis, prognosis and treatment. Neurol Clin. 2011 Nov;29(4):773-86. doi: 10.1016/j.ncl.2011.07.009. PMID 22032660
- [Background] Laureys S, Owen AM, Schiff ND. Brain function in coma, vegetative state, and related disorders. Lancet Neurol. 2004 Sep;3(9):537-46. doi: 10.1016/S1474-4422(04)00852-X. PMID 15324722
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Bruno MA, Vanhaudenhuyse A, Thibaut A, Moonen G, Laureys S. From unresponsive wakefulness to minimally conscious PLUS and functional locked-in syndromes: recent advances in our understanding of disorders of consciousness. J Neurol. 2011 Jul;258(7):1373-84. doi: 10.1007/s00415-011-6114-x. Epub 2011 Jun 16. PMID 21674197
- [Background] Calabro RS, Naro A. Diagnosing Disorder of Consciousness: The Opening of Pandora's Box! Innov Clin Neurosci. 2016 Apr 1;13(3-4):10-1. eCollection 2016 Mar-Apr. No abstract available. PMID 27354922
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] 'CRSR_GeneralGuidelines_20200812_v1.pdf'. Accessed: Jun. 09, 2022. [Online]. Available: https://www.sralab.org/sites/default/files/downloads/2020-09/CRSR_GeneralGuidelines_20200812_v1.pdf
- [Background] J. T. Giacino, 'COMA RECOVERY SCALE-REVISED ©2004', p. 17, 2020.
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] American Congress of Rehabilitation Medicine, Brain Injury-Interdisciplinary Special Interest Group, Disorders of Consciousness Task Force; Seel RT, Sherer M, Whyte J, Katz DI, Giacino JT, Rosenbaum AM, Hammond FM, Kalmar K, Pape TL, Zafonte R, Biester RC, Kaelin D, Kean J, Zasler N. Assessment scales for disorders of consciousness: evidence-based recommendations for clinical practice and research. Arch Phys Med Rehabil. 2010 Dec;91(12):1795-813. doi: 10.1016/j.apmr.2010.07.218. PMID 21112421
- [Background] Gerrard P, Zafonte R, Giacino JT. Coma Recovery Scale-Revised: evidentiary support for hierarchical grading of level of consciousness. Arch Phys Med Rehabil. 2014 Dec;95(12):2335-41. doi: 10.1016/j.apmr.2014.06.018. Epub 2014 Jul 7. PMID 25010536
- [Background] La Porta F, Caselli S, Ianes AB, Cameli O, Lino M, Piperno R, Sighinolfi A, Lombardi F, Tennant A. Can we scientifically and reliably measure the level of consciousness in vegetative and minimally conscious States? Rasch analysis of the coma recovery scale-revised. Arch Phys Med Rehabil. 2013 Mar;94(3):527-535.e1. doi: 10.1016/j.apmr.2012.09.035. Epub 2012 Nov 2. PMID 23127303
- [Background] Schnakers C, Vanhaudenhuyse A, Giacino J, Ventura M, Boly M, Majerus S, Moonen G, Laureys S. Diagnostic accuracy of the vegetative and minimally conscious state: clinical consensus versus standardized neurobehavioral assessment. BMC Neurol. 2009 Jul 21;9:35. doi: 10.1186/1471-2377-9-35. PMID 19622138
- [Background] Wannez S, Heine L, Thonnard M, Gosseries O, Laureys S; Coma Science Group collaborators. The repetition of behavioral assessments in diagnosis of disorders of consciousness. Ann Neurol. 2017 Jun;81(6):883-889. doi: 10.1002/ana.24962. PMID 28543735
- [Background] Jox RJ, Bernat JL, Laureys S, Racine E. Disorders of consciousness: responding to requests for novel diagnostic and therapeutic interventions. Lancet Neurol. 2012 Aug;11(8):732-8. doi: 10.1016/S1474-4422(12)70154-0. PMID 22814543
- [Background] Sattin D, Minati L, Rossi D, Covelli V, Giovannetti AM, Rosazza C, Bersano A, Nigri A, Leonardi M. The Coma Recovery Scale Modified Score: a new scoring system for the Coma Recovery Scale-revised for assessment of patients with disorders of consciousness. Int J Rehabil Res. 2015 Dec;38(4):350-6. doi: 10.1097/MRR.0000000000000135. PMID 26465775
- [Background] Annen J, Filippini MM, Bonin E, Cassol H, Aubinet C, Carriere M, Gosseries O, Thibaut A, Barra A, Wolff A, Sanz LRD, Martial C, Laureys S, Chatelle C. Diagnostic accuracy of the CRS-R index in patients with disorders of consciousness. Brain Inj. 2019;33(11):1409-1412. doi: 10.1080/02699052.2019.1644376. Epub 2019 Jul 18. PMID 31319707
- [Background] Estraneo A, Moretta P, Loreto V, Lanzillo B, Cozzolino A, Saltalamacchia A, Lullo F, Santoro L, Trojano L. Predictors of recovery of responsiveness in prolonged anoxic vegetative state. Neurology. 2013 Jan 29;80(5):464-70. doi: 10.1212/WNL.0b013e31827f0f31. Epub 2013 Jan 9. PMID 23303855
- [Background] Practice Guideline Update Recommendations Summary_ Disorders of Consciousness.pdf'.
- [Background] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Practice guideline update recommendations summary: Disorders of consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Neurology. 2018 Sep 4;91(10):450-460. doi: 10.1212/WNL.0000000000005926. Epub 2018 Aug 8. PMID 30089618
- [Background] Martens G, Bodien Y, Sheau K, Christoforou A, Giacino JT. Which behaviours are first to emerge during recovery of consciousness after severe brain injury? Ann Phys Rehabil Med. 2020 Jul;63(4):263-269. doi: 10.1016/j.rehab.2019.10.004. Epub 2019 Nov 26. PMID 31783144
- [Background] Carriere M, Llorens R, Navarro MD, Olaya J, Ferri J, Noe E. Behavioral signs of recovery from unresponsive wakefulness syndrome to emergence of minimally conscious state after severe brain injury. Ann Phys Rehabil Med. 2022 Mar;65(2):101534. doi: 10.1016/j.rehab.2021.101534. Epub 2021 Nov 18. PMID 33933691
- [Background] Liuzzi P, Grippo A, Campagnini S, Scarpino M, Draghi F, Romoli A, Bahia H, Sterpu R, Maiorelli A, Macchi C, Cecchi F, Carrozza MC, Mannini A. Merging Clinical and EEG Biomarkers in an Elastic-Net Regression for Disorder of Consciousness Prognosis Prediction. IEEE Trans Neural Syst Rehabil Eng. 2022;30:1504-1513. doi: 10.1109/TNSRE.2022.3178801. Epub 2022 Jun 13. PMID 35635833
- [Background] Noe E, Ferri J, Olaya J, Navarro MD, O'Valle M, Colomer C, Moliner B, Ippoliti C, Maza A, Llorens R. When, How, and to What Extent Are Individuals with Unresponsive Wakefulness Syndrome Able to Progress? Neurobehavioral Progress. Brain Sci. 2021 Jan 19;11(1):126. doi: 10.3390/brainsci11010126. PMID 33478033
- [Background] Arnaldi D, Terzaghi M, Cremascoli R, De Carli F, Maggioni G, Pistarini C, Nobili F, Moglia A, Manni R. The prognostic value of sleep patterns in disorders of consciousness in the sub-acute phase. Clin Neurophysiol. 2016 Feb;127(2):1445-1451. doi: 10.1016/j.clinph.2015.10.042. Epub 2015 Nov 6. PMID 26610323
- [Background] Magliacano A, Liuzzi P, Formisano R, Grippo A, Angelakis E, Thibaut A, Gosseries O, Lamberti G, Noe E, Bagnato S, Edlow BL, Lejeune N, Veeramuthu V, Trojano L, Zasler N, Schnakers C, Bartolo M, Mannini A, Estraneo A; IBIA DoC-SIG. Predicting Long-Term Recovery of Consciousness in Prolonged Disorders of Consciousness Based on Coma Recovery Scale-Revised Subscores: Validation of a Machine Learning-Based Prognostic Index. Brain Sci. 2022 Dec 27;13(1):51. doi: 10.3390/brainsci13010051. PMID 36672033